CLINICAL TRIAL: NCT04200495
Title: PSG Validation Study of Zensorium Biosensing Wearable Device
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: Nitto Denko Asia Technical Centre (NAT) (Unknown)
Responsible Party: Principal Investigator, Peter Colvonen, Assistant Clinical Professor, University of California, San Diego
Other Study IDs: 190705
Record Dates: First submitted 2019-12-06; First posted 2019-12-16 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Sleep Wake Disorders; Healthy
MeSH Terms: conditions — Sleep Wake Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Controls: No sleep-wake disorder present
- Active Sleep-Wake Disorder: Presence of Sleep-Wake Disorder

SUMMARY:
The objective of this study is to collect data comparing the Zensorium Biosensing Wearable Device (zBWD) to polysomnography (PSG) in individuals with Sleep-Wake Disorders. zBWD is similar to other wearable devices (e.g., fitbit and apple watch) that use an optical light sensor and Tri-axis Accelerometer to record steps, activity, sleep/awake states, sleep staging, and statistical variation of pulse pressure to track stress. Specifically, it is designed to report sleep duration, non-rapid eye movement (NREM) and REM sleep duration. However, zBWD has not been validated against PSG for sleep tracking in healthy controls or in individuals with sleep-wake disorders.

DETAILED DESCRIPTION:
Subjects known to have or not have sleep-wake disorder, as well as healthy subjects, will be enrolled if they otherwise meet all the inclusion criteria, and none of the exclusion criteria. Subject will be asked to complete several questionnaires and wear the zBWD for 7-days, in an off-site (Home) study, followed by a single overnight PSG study to compare the zBWD data to the current gold standard of PSG. Subjects who have completed the study will also be sent a letter thanking them for their participation and offering a summary of the results of their sleep study.

ELIGIBILITY:
Inclusion Criteria:

* 1. Health status: Healthy, or those with sleep-wake disorders

Exclusion Criteria:

1. Pregnancy
2. Currently smoking
3. Any respiratory disorder other than associated with Sleep/Wake Disorder or well-controlled asthma
4. Habitual use of medications known to affect respiratory function (e.g. opioids, benzodiazepines, etc).
5. Use of medication known to affect pulse pressure (Beta Blockers)
6. Atrial Fibrillation
7. Tattoos located on wrist

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Healthy adults and those with sleep/Wake Disorders
Sampling Method: Non-Probability Sample
Enrollment: 68 (Actual)
Dates: Start 2019-11-20 (Actual); Primary Completion 2020-10-28 (Actual); Study Completion 2020-10-28 (Actual)

PRIMARY OUTCOMES:
polysomnography derived percent REM and percent non-REM sleep | One overnight stay at Visit 2 (7 - 10 days following Baseline)
  A full clinical overnight polysomnography (PSG) study will be performed 7 - 10 days following visit 1. The subject will have EEG, EMG, EOG, and ECG electrodes, an adhesive body position sensor placed in standard locations. This equipment is standard for diagnostic PSG. The variables of interest from the PSG are stages of sleep as indicated by PSG including % rapid eye movement (REM; amount of time in REM sleep/Total sleep time) and % non-REM (amount of time in non-REM sleep/Total sleep time)
Zensorium derived percent REM and percent Non-REM sleep | To be worn everyday between Baseline to visit 2 (7 -10 days)
  Zensorium Biosensing Wearable Device (zBWD) will be worn for 7 to 10 days following visit 1. The variables of interest are stages of sleep as indicated by the zBWD including % rapid eye movement (REM; amount of time in REM sleep/Total sleep time) and % non-REM (amount of time in non-REM sleep/Total sleep time).

SECONDARY OUTCOMES:
Sleep Diary | To be filled out everyday between Baseline to visit 2 (7 -10 days)
  Tracking off-site (home) sleep for 7 to 10 days via self report diary - Sleep Efficiency, Total Sleep Time, Sleep latency, and Wake after sleep onset
Insomnia Severity Index | Baseline
  Insomnia Severity Index (ISI) is a widely used measure of insomnia with well-established reliability and validity. The ISI consists of seven items, three of which assess severity of insomnia (i.e., degree of difficulty falling asleep, staying asleep, and waking too early). The remaining questions tap satisfaction with sleep pattern, effect of sleep on daytime and social functioning, and concern about current sleep difficulties. Ranges from 0 (no insomnia) to 28 (Severe insomnia)
Pre-Sleep Arousal Scale | Baseline
  Pre-sleep arousal scale (PSAS) is a self-administered measure in which participants rate the intensity of experienced arousal for somatic (8 items) and cognitive (8 items) subscales. The PSAS shows strong internal consistency and reliability. Higher scores indicate worse pre-sleep arousal. Ratings range from 1 (not at all) to 5 (extremely).
Berlin Questionnaire | Baseline
  Berlin Questionnaire is a validated screening tool for sleep disordered breather. One question and four follow-up questions concern snoring; three questions address daytime sleepiness, with a subquestion about sleepiness behind the wheel. Lastly, the measure addresses history of high blood pressure, age, weight, height, sex, neck circumference, and ethnicity. High Risk is considered if there are 2 or more categories where the score is positive, where more categories endorsed equates to higher risk.
Epworth Sleepiness Scale | Baseline
  Epworth Sleepiness Scale (ESS) is a self-administered questionnaire with 8 questions. The questions measure participants experiences of having dozed off or fallen asleep while engaged in eight different activities that differ widely in their somnificity (including sitting in traffic or watching television). can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No